CLINICAL TRIAL: NCT02236715
Title: Postmarketing Surveillance Study (as Per §67(6)AMG[German Drug Law]) of Atrovent® Unit Dose Vial 500 µg in Chronic Obstructive Airways Disease
Brief Title: Postmarketing Surveillance Study of Atrovent® in Chronic Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 244.2493
Record Dates: First submitted 2014-09-10; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ipratropium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Obstructive Airways Disease
  Interventions: Drug: Atrovent®

INTERVENTIONS:
Drug: Atrovent®

SUMMARY:
Study to obtain further information on the tolerability and efficacy of Atrovent® unit dose vial 500 µg in the treatment of Chronic Obstructive Airways Disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Primarily patients of both gender, older than 30 years, who suffer from chronic obstructive airways disease
* Only patients who had not been treated with Atrovent® within the last year were to be considered for inclusion

Exclusion Criteria:

* Contraindication listed in the instructions for use/summary of product characteristics for Atrovent® unit dose vial 500 µg

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive airways disease recruited at general practitioners, pneumologists, internists
Sampling Method: Non-Probability Sample
Enrollment: 1039 (Actual)
Dates: Start 1999-09; Primary Completion 2000-02 (Actual)

PRIMARY OUTCOMES:
Change in total severity of the clinical picture rated on a 4-point scale | after 4 weeks

SECONDARY OUTCOMES:
Assessment of efficacy by investigator on a 4-point scale | after 4 weeks
Assessment of efficacy by patient on a 4-point scale | after 4 weeks
Assessment of tolerability by investigator on a 4-point scale | after 4 weeks
Assessment of tolerability by patient on a 4-point scale | after 4 weeks
Number of patients with adverse drug reactions | up to 4 weeks